CLINICAL TRIAL: NCT01379014
Title: The CORAL Study of a Decision Aid Tool Regarding Disclosure of Mental Health Status to an Employer: Proof of Concept Randomised Control Trial
Brief Title: CORAL Study: Proof of Concept Trial
Acronym: CORAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Psychiatry, London (Other)
Responsible Party: Principal Investigator, Claire Henderson, MRCPsych MSc PhD, Dr Claire Henderson, Institute of Psychiatry, London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 11/EE/0156
Record Dates: First submitted 2011-06-17; First posted 2011-06-23 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Mental Illness
Keywords: Decisional conflict; Disclosure; Mental Health history; Mental health service users; Decision Aid Tool; Vocational Specialists
MeSH Terms: conditions — Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Aid Tool (Experimental): Intervention group - receives the decision aid tool in booklet form and is introduced to it by an investigator.
  Interventions: Behavioral: Decision Aid Tool
- Control (No Intervention): The control group does not receive a copy of the decision aid tool booklet, instead received treatment as usual from vocational specialist
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Decision Aid Tool — A booklet which outlines to pros and cons of different decision outcomes, and is designed to assist the user in making a decision according to their own specific circumstances
  Arms: Decision Aid Tool
Other: Treatment as Usual — The control group does not receive a copy of the decision aid tool booklet, instead received treatment as usual from vocational specialist
  Arms: Control

SUMMARY:
A decision aid tool (DAT) to assist mental health service users in reaching disclosure decisions in the context of employment was developed in a previous study (IRAS REC ref: 07/Q0706/21). The initial feasibility and acceptability was assessed in a group of 15 mental health service users with mean decisional conflict scores reduced from 51.98 to 35.52 after completion. 60% of participants reported that the DAT was quick to complete, 40% that it was easy, 60% that it was relevant and 80% that they would definitely or probably use it in making disclosure decisions. This current study (CORAL: Proof of concept RCT) aims to determine whether a full randomised controlled trial of the DAT is justifiable and feasible, and to optimise its design. This will consider: 1) effects of the intervention; 2) baseline predictors of disclosure; and 3) exploration of the relationship between use of the DAT and the rate of disclosure.

Eighty people who are on the caseload of a vocational specialist working with people with mental illness will be included in this study. All participants will be receiving treatment from an Improving Access to Psychological Therapies (IAPT) service or a Community Mental Health Team (CMHT). An equal number from each group will be allocated to receive either the DAT intervention or treatment as usual. Individuals from both groups will complete baseline assessment and 3month followup assessments. Those allocated to the intervention will also complete an assessment immediately following the intervention. Qualitative interviews will also be conducted at 3 months with a maximum of 15 people from the intervention group and 6 people from the control group.

DETAILED DESCRIPTION:
The principal aims are to determine whether a full randomised controlled trial of the CORAL decision aid tool is justifiable and feasible and to optimise its design. Specific objectives are as follows:

1. To examine the effect of the DAT on decisional conflict regarding disclosure both immediately and at 3 months post first use.
2. To collect data to inform sample size calculations for the primary outcome measures for use in a future full scale trial(gaining employment and workplace accommodations).
3. To test study procedures, including the sample that can be drawn using the inclusion and exclusion criteria; the full time equivalent needed for research assistants to recruit sufficient numbers and carry out the study procedures in the time available; and whether the measure leads to too much respondent burden.
4. To pilot the use of a questionnaire on employment and disclosure related activities.
5. To test the selected randomisation method, in this case individual level randomisation, including the methods for avoiding and measuring contamination.
6. To pilot recruitment and retention methods for service users and vocational specialists.
7. To estimate effect sizes and their confidence intervals for employment related activities (proxy outcome measures for gaining employment and workplace accommodations), in order to determine whether a full scale trial is justified.
8. To modify the conceptual model

ELIGIBILITY:
Inclusion Criteria:

1. On the caseload of a vocational specialist working with people with mental illness.
2. Referred to the adviser either from an Increased Access to Psychological Therapies or secondary mental health care service.
3. Aged 18 years or older
4. Currently seeking either paid or voluntary employment or interested in seeking paid or voluntary employment
5. Decisional conflict scale score of 37.5 or greater and stage of decision score 1-5

Exclusion Criteria:

1. Insufficient English to use the decision aid tool
2. Lack of capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
decisional conflict scale | Change from baseline in decisional conflict at 3 months
  Decisional conflict scale (O'Connor, 1993) This measures personal perceptions of uncertainty, lack of clarity and effectiveness in decision making. Has 16 items with each rated on a 5 point Likert scale ranging from 0=strongly agree to 4=strongly disagree.

SECONDARY OUTCOMES:
Sociodemographic data | baseline
  Socio-demographic and clinical data to be collected as part of the baseline interview will include age, gender, years since first contact with mental health services, education, employment status and history, housing arrangements, source of income, current mental health care, knowledge of clinical diagnosis, agreement with diagnosis and information on social networks.
Employment related questions | baseline and 3-month follow up
  To record how many jobs applications, apppointments with vocational specialists, training days and job applications the participant has completed in the preceeding 3 months.
Discrimination and Stigma Scale (DISC) | Baseline and 3-month follow-up
  scale to assess mental health service users' experiences of discrimination. 22 items. Baseline assesses if discrimination/stigma has ever been experienced, 3 month follow-up asks if discrimination/stigma as been experienced in the past three months.
  Thornicroft, G., Brohan, E., Rose, D., Sartorius, N. & the INDIGO study group. (2009) Global pattern of experienced and anticipated discrimination against people with schizophrenia. The Lancet, 373 (9661), 408-415
Questionnaire on Anticipated Discrimination (QUAD) | baseline and 3 month follow-up
  The QUAD is a self-complete measure which contains 17 items which address 'areas of anticipated discrimination'. This asks participants to provide a rating of whether they expect to be treated unfairly in various areas of life. Each item is scored on a five point Likert scale ranging from 0 (Strongly disagree) to 4 (Strongly agree).
  Brohan E, Clement S, Thornicroft G. Development and initial validation of the questionnaire on anticipated discrimination (QUAD v6, May 2011) © 2011, Institute of Psychiatry, King's College London
Boston University Empowerment Scale (BUES) | baseline and 3 month follow-up
  This 28-item scale was developed with an emphasis on service user-involvement at all stages of design and testing. This version has shown adequate internal consistency (α=.86).
  Rogers, E. S., Chamberlin, J., Ellison, M. L., et al (1997) A consumer-constructed scale to measure empowerment among users of mental health services. Psychiatric Services, 48, 1042-1047.
Internalised Stigma of Mental Illness Scale (ISMI) | Baseline and 3 month follow-up
  The ISMI is a 29-item measure that assesses mental health service users' experience of internalised stigma. It is composed of 5 sub-scales: Alienation, Stereotype Endorsement, Perceived Discrimination, Social Withdrawal and Stigma Resistance. Strong internal consistency (α = 0.90) and test-retest reliability(r=0.92) have been reported Ritsher JB, Otilingam PG, Grajales M. Internalized stigma of mental illness: Psychometric properties of a new measure. Psychiatry Research 2003;121(1):31-49.
Perceived Devaluation and Discrimination Scale (PDD) | Baseline and 3 month follow-up
  The PDD is a 12-item, uni-dimensional, scale which measures the extent to which a person believes that people will devalue or discriminate against those with a mental illness. This scale has been widely used and has excellent psychometric properties
  Link, B.G., Neese-Todd, S., Asmussen, S. & Phelan, J.C. (2002). On describing and seeking to change the experience of stigma. Psychiatric Rehabilitation Skills, 6: 201-231.
Stigma Coping Orientation Scales | baseline and 3 month follow-up
  Measures to assess approaches to coping with the stigma associated with mental illness. Revised versions of four of the scales are now available and will be used in this study. These are secrecy (5-items alpha = .85), withdrawal (5-items alpha = .71), challenging (5 items alpha = .75) and distancing (3 items alpha = .62) (Bruce Link, personal communication).
  The Effectiveness of Stigma Coping Orientations: Can Negative Consequences of Mental Illness Labeling be Avoided? Bruce G. Link, Jerrold Mirotznik, Francis T. Cullen, Journal of Health and Social Behavior, Vol. 32, No. 3 (Sep., 1991)
Brief COPE | Baseline and 3-months Follow-up
  A short-version COPE Inventory. Assesses response to stress. 14 scales with two items each; self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion and self-blame. Reliability analyses exceeded alpha=0.60, except for venting, denial and acceptance, all of which exceed alpha = 0.50 (Carver et al 1997)
  Carver, C. S. (1997). International Journal of Behavioral Medicine, 4, 92-100
Work Limitations Questionnaire (WLQ) | Baseline and 3 month follow-up (for those in employment only)
  The 8-item short WLQ measures the degree to which employed individuals are experiencing limitations on-the-job due to their health problems, and health-related productivity loss.
  Work Limitations Questionnaire, 1998. The Health Institute, Tufts Medical Center, 800 Washington Street, Nemc #345, Boston, MA 02111
stage of decision making scale | Baseline and 3 month follow-up
  Stage of decision making scale (O'Connor, 2000).This measures the individual's readiness to engage in decision making It consists of 1 item with 6 response options anchored at 1 (haven't started to think about the choices) and 6 (have already made a decision and am unlikely to change my mind).

CONTACTS AND LOCATIONS:
Overall Officials: Graham Thornicroft, FRCPsych, Study Director — Institute of Psychiatry, London
Locations (1):
- Institute of Psychiatry, King's College London, London, United Kingdom

REFERENCES:
- [Derived] Henderson C, Brohan E, Clement S, Williams P, Lassman F, Schauman O, Dockery L, Farrelly S, Murray J, Murphy C, Slade M, Thornicroft G. Decision aid on disclosure of mental health status to an employer: feasibility and outcomes of a randomised controlled trial. Br J Psychiatry. 2013 Nov;203(5):350-7. doi: 10.1192/bjp.bp.113.128470. Epub 2013 Sep 26. PMID 24072755
- [Derived] Henderson C, Brohan E, Clement S, Williams P, Lassman F, Schauman O, Murray J, Murphy C, Slade M, Thornicroft G. A decision aid to assist decisions on disclosure of mental health status to an employer: protocol for the CORAL exploratory randomised controlled trial. BMC Psychiatry. 2012 Aug 31;12:133. doi: 10.1186/1471-244X-12-133. PMID 22938019
- See also: Institute of Psychiatry homepage — http://www.kcl.ac.uk/iop/index.aspx